CLINICAL TRIAL: NCT01093989
Title: Acute vs. Delayed Iron Therapy: Effect on Iron Status, Anemia and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0909M72852; 1U01HD064698-01 (NIH)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Anemia; Inflammation; Malaria Morbidity; Cognitive Development
MeSH Terms: conditions — Anemia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate iron (Placebo Comparator): Iron-deficient children will be randomized to receive iron concurrently with anti-malarial treatment or one month later (delayed iron group).
  Interventions: Dietary Supplement: Ferrous Sulphate Syrup
- Delayed iron (Active Comparator)
  Interventions: Dietary Supplement: Ferrous Sulphate Syrup

INTERVENTIONS:
Dietary Supplement: Ferrous Sulphate Syrup — Iron therapy will consist of a three-month course of ferrous sulphate syrup. For children with Hb ≥ 7 g/dL, each daily dose will be based on 2 mg iron/kg body weight.

SUMMARY:
The research questions to be answered by this study are:

1. Is treatment with iron more effective at improving anemia if given at the time of a malaria episode or 1 month after the episode?
2. Which treatment timing is associated with more malaria episodes - 1 month delayed treatment or immediate treatment at the time of malaria?
3. Does timing of iron treatment affect later thinking processes and behavior?

DETAILED DESCRIPTION:
The study population in this study will be children who are enrolled in our ongoing study of cerebral malaria and severe malarial anemia, "Pathogenesis of cognitive/neurologic deficits in central nervous system malaria", underway in Kampala, Uganda. The pathogenesis study seeks to address the question of why children with severe malaria have later problems in thinking. The study we are now proposing will build on this study by assessing whether children with severe malaria have iron deficiency, and if they do, whether treatment with iron at the time of malaria is less effective than treatment one month later. We believe that treatment one month later may be more effective because there is data that shows that the inflammation that occurs with a malaria episode may decrease the body's ability to absorb iron in the gut and to send iron to the places it is needed, like the bone marrow and the brain. We are doing this study to see if our hypothesis about more effective iron treatment if it is delayed is correct and assessing anemia prevalence, iron status, and long-term neurobehavioral development as outcomes.

We have three study groups: children with cerebral malaria, children with severe malarial anemia, and healthy community control children. Children found to be iron deficient will be randomized to receive iron (as ferrous sulphate syrup) either immediately or at their one-month follow-up visit. At 1-, 6, and 12-month follow-up visits changes in iron and inflammation indicators will be assessed. At the 6- and 12-month visits, neurocognitive behavior will also be evaluated and compared between the immediate vs. delayed iron groups. Malaria morbidity will be assessed via home visits during the period of iron supplementation and via clinic monitoring for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* All children must

  1. Be between the ages of 18 mo and 5 y
  2. Reside within 20 km of study hospital
* Children with cerebral malaria must have

  1. Coma (BCS < 3)
  2. P. falciparum on blood smear
  3. No clinical evidence or other causes of encephalopathy
* Children with severe malarial anemia must have

  1. Hemoglobin < 5 g/dL
  2. Clinical symptoms of malaria
  3. P. falciparum on blood smear
* Community control children must

  1. Live in same neighborhood or extended household as a child with severe malaria
  2. Be within one year of age as a child with severe malaria

Exclusion Criteria:

* Cerebral malaria

  1. WBC > 10
  2. Positive gram stain or culture

Severe malarial anemia

1. Impaired conscious on physical exam
2. Seizure activity prior to or during physical exam
3. Any other evidence of CNS disease
4. All exclusion criteria of CM except no lumbar puncture required

Community control children

1. All exclusion criteria for CM
2. Any active illness, recent illness, or recovery from illness
3. Chronic illness requiring medical care
4. Medical abnormalities on screening history of physical exam
5. CC control with a positive malaria smear will be treated but will not be excluded from the study.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin change, anemia prevalence, and socioemotional behavior in the immediate iron vs. delayed iron groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C John, M.D., Principal Investigator — University of Minnesota
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Blatt DB, Hanisch B, Co K, Datta D, Bond C, Opoka RO, Cusick SE, Michelow IC, John CC. Impact of Oxidative Stress on Risk of Death and Readmission in African Children With Severe Malaria: A Prospective Observational Study. J Infect Dis. 2022 Sep 4;226(4):714-722. doi: 10.1093/infdis/jiac234. PMID 35678643
- [Derived] Cusick SE, Opoka RO, Ssemata AS, Georgieff MK, John CC. Delayed iron improves iron status without altering malaria risk in severe malarial anemia. Am J Clin Nutr. 2020 May 1;111(5):1059-1067. doi: 10.1093/ajcn/nqaa004. PMID 32005992
- [Derived] Cusick SE, Opoka RO, Ssemata AS, Georgieff MK, John CC. Comparison of iron status 28 d after provision of antimalarial treatment with iron therapy compared with antimalarial treatment alone in Ugandan children with severe malaria. Am J Clin Nutr. 2016 Mar;103(3):919-25. doi: 10.3945/ajcn.115.117820. Epub 2016 Feb 3. PMID 26843153